CLINICAL TRIAL: NCT02755155
Title: Comparison of 2 Strategies of Therapeutic Human Serum Albumin Infusion in Critically Ill Patients With Severe Systemic Inflammatory Response Syndrome and Low Plasma Albumin: Continuous Low Versus Intermittent High Doses
Brief Title: Optimization of Therapeutic Human Serum Albumin Infusion in Selected Critically Ill Patients
Acronym: AlbAlsace
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: too many patients were expected and the investigative team would not be able to recruit this number
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6371
Record Dates: First submitted 2016-04-13; First posted 2016-04-28 (Estimated); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Shock; Systemic Inflammatory Response Syndrome (SIRS); Hypoalbuminaemia
Keywords: acute circulatory failure requiring norepinephrine; SIRS; Albumin, therapeutic
MeSH Terms: conditions — Shock; Systemic Inflammatory Response Syndrome; Hypoalbuminemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous low dosage (CLD) (Experimental): The subjects will received human serum albumin infusion 4%.CLD patients are infused with15ml/kg/day of 4% human serum albumin from inclusion to the day norepinephrine infusion is weaned by 30% (provided their plasma albumin stays in the range 30+3g/L)
  Interventions: Drug: Human serum albumin infusion 4%
- Intermittent high dosage (IHD) (Active Comparator): The subjects will received human serum albumin infusion 20%.IHD patients are infused with 20% human serum albumin (up to 600 ml/day) until the plasma albumin concentration is in the range 30+3g/L from inclusion to the day norepinephrine infusion is weaned by 30%
  Interventions: Drug: Human serum albumin infusion 20%

INTERVENTIONS:
Drug: Human serum albumin infusion 4% — Continuous infusion of 15mL/kg of bodyweight over 24h/day
  Other Names: VIALEBEX* 4%
  Arms: Continuous low dosage (CLD)
Drug: Human serum albumin infusion 20% — Specify details not covered in associated Arm Description. Intermittent infusion up to 200 ml/8h/day until the plasma albumin concentration is in the range 30+3g/L
  Other Names: VIALEBEX* 20%
  Arms: Intermittent high dosage (IHD)

SUMMARY:
Primary purpose : mortality at Day 28

Secondary purposes :

* Daily SOFA (Sequential Organ Failure Assessment) score lessening within Intensive Care Unit (ICU)
* Duration of increasing doses of norepinephrine infusion to maintain target mean arterial pressure
* Number of care-related infections within ICU

DETAILED DESCRIPTION:
According to currently available literature on therapeutic albumin infusion in critically ill patients, there is room for new approaches to delineate an optimal use of this expansive treatment. Indeed, many authors suggest that the present clinical use of albumin is questionable in critically ill patients as far as changes in morbidity or mortality are concerned and with regards to cost-effectiveness.

It has been reported that protein misfolding and aggregation are a hallmark of several inflammatory diseases. In vitro studies show that very small amounts of albumin are able to restore the physiologic activities of endogenous circulating proteins that had been aggregated in multimeric form during oxidative stress. Recently, the investigators have reported that in vitro albumin restores antimicrobial and anti-inflammatory effects of some chromogranin A-derived peptides. The investigators therefore search to test in vivo, in critically ill patients with severe systemic inflammation requiring norepinephrine infusion, whether therapeutic albumin infused at a low and continuous dosage may modify mortality (primary purpose) and morbidity (secondary purposes) in comparison with intermittent high dosage albumin infusion.

ELIGIBILITY:
Inclusion Criteria:

* circulatory failure requiring norepinephrine support (any dose)
* hospitalization within an Intensive Care Unit
* SIRS
* low plasma albumin (< 20g/L)
* consent to study

Exclusion Criteria:

* absence of circulatory failure
* absence of SIRS
* chronic low albumin concentration
* absence of consent to study
* inability to tolerate human serum albumin
* Patients under guardianship or curators
* Women pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2019-08-10 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 days after inclusion between the two groups

SECONDARY OUTCOMES:
The length of the circulatory failure requiring albumin infusion | The estimated period of time will be from date of baseline visit until the date of discharge from the hospital or date of death from any cause, whichever came first, assessed up to 28 days
  Time from albumin infusion starting to the moment when norepinephrine can be weaned at least by 30% of its peak dose with respect of initial mean arterial pressure target between the two groups.

OTHER OUTCOMES:
Daily SOFA score | The outcome measure will be assessed from date of baseline visit until the date of discharge from the hospital or date of death from any cause, whichever came first, assessed up to 28 days
  Daily SOFA score decrease from albumin infusion starting to norepinephrine weaning at least by 30% of its peak dose between the two groups
The number of infections in intensive care | Number of care-related infection within intensive care (28 days) unit between the two groups.
  The outcome will be assessed with the adverse event notification

CONTACTS AND LOCATIONS:
Overall Officials: Francis SCHNEIDER, Prof, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaire de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No